CLINICAL TRIAL: NCT06885086
Title: The Impact of ERAS-Based Multimodal Pain Management on Clinical Outcomes in Laparoscopic Cholecystectomy: Ambispective Cohort Study
Brief Title: ERAS (Enhanced Recovery After Surgery) and Multimodal Analgesia in Laparoscopic Cholecystectomy
Acronym: ERAS
Status: Not yet recruiting | Type: Observational
Sponsor: Cukurova University (Other)
Collaborators: Toros University (Other)
Responsible Party: Principal Investigator, Esma Gökçe, Assistant Professor, Cukurova University
Other Study IDs: ERAS-LC-2025
Record Dates: First submitted 2025-03-07; First posted 2025-03-20 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Pain Management; Cholecystectomy, Laparoscopic; Perioperative Care; Analgesia; Surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group - 1: In the control group (previous standard care), no analgesic was administered intraoperatively. Postoperative analgesia was provided on an as-needed basis according to patients' pain levels. Accordingly, intravenous paracetamol (1 g, three times daily), intramuscular NSAIDs (twice daily), and intravenous opioids (tramadol; 50/100 mg once daily, based on patient weight) were prescribed pro re nata (PRN). These medications were not given routinely but only when a significant increase in pain was observed. The data required for the control group-including analgesic doses and information from data collection forms-will be obtained retrospectively from archive records.
  Interventions: Other: Control group - 1
- Observation group -2: Thirty minutes before anesthesia induction, 1 g of intravenous paracetamol is administered. During the intraoperative period, prior to wound closure, 800 mg of intravenous ibuprofen (diluted in 250 mL of normal saline) is administered. After trocar removal, 10 mL of 0.5% bupivacaine is infiltrated subcutaneously into the surgical wounds.
  Postoperatively, patients receive oral paracetamol (1 g every 6 hours) and oral ibuprofen (400 mg every 8 hours). If the Visual Analog Scale (VAS) score exceeds 7, an additional opioid intervention is provided using oral Contramal (tramadol) (50/100 mg, based on patient weight).
  For the observation group, a preoperative sociodemographic form is completed, and the VAS pain score is recorded at 2, 4, 8, 12, 18, and 24 hours postoperatively. Additionally, a clinical information and complication form is filled out before discharge.
  Interventions: Drug: Observation group -2

INTERVENTIONS:
Other: Control group - 1 — Patient data will be collected retrospectively from the records.
  Other Names: Retrospective group
  Groups: Control group - 1
Drug: Observation group -2 — In the literature, multimodal analgesia strategies-as recommended by ERAS guidelines and supported by recent studies-are implemented. In the intraoperative period, patients receive paracetamol, NSAIDs, and local surgical wound infiltration analgesia. In the postoperative period, oral paracetamol and NSAIDs are routinely continued, with opioids administered as needed.
  Other Names: Prospective group
  Groups: Observation group -2

SUMMARY:
This clinical study aims to evaluate the effects of multimodal analgesia management administered within an ERAS (Enhanced Recovery After Surgery) protocol on postoperative pain, length of hospital stay, early complications, and additional opioid requirements in patients undergoing laparoscopic cholecystectomy. The key questions addressed are:

* Does ERAS-based multimodal analgesia reduce postoperative pain?
* Does it shorten the hospital stay and lower early complication rates?
* What is its potential to reduce the need for additional opioids?

Participants:

* Prospective Group: Patients managed with an ERAS multimodal analgesia protocol (including paracetamol, NSAIDs (Non-Steroidal Anti-Inflammatory Drugs), and local wound infiltration analgesics) between April and July 2025.
* Retrospective Group: Patient records from 2024 who were treated with a routine analgesia protocol.

Based on a power analysis, a minimum of 60 patients per group (total of 120 patients) will be included in the study (If the required sample size determined by the power analysis cannot be reached, the number of patients within the predefined time frame will be accepted as the sample).

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy is regarded as the gold standard minimally invasive surgical method for treating gallstones and cholecystitis. This approach offers significant advantages over open surgery, including lower complication rates, shorter hospital stays, and faster postoperative recovery. Nevertheless, postoperative recovery and the risk of complications remain important concerns.

The Enhanced Recovery After Surgery (ERAS) protocol is a comprehensive approach developed to accelerate postoperative recovery and reduce complications. It includes numerous components applied during the preoperative, intraoperative, and postoperative periods, all aiming to shorten recovery time and enhance patient comfort.

A key element of ERAS protocols in surgical practice is pain management. Postoperative pain directly affects both the psychological and physiological recovery of surgical patients and is a critical clinical issue regarding treatment response and quality of life. Inadequate pain control may lead to delayed early mobilization, prolonged hospital stays, the development of chronic pain, and an increased risk of side effects associated with heightened opioid use. The concurrent use of multiple analgesic drugs or techniques, each targeting different pain mechanisms, has been advocated to reduce opioid-related side effects while enhancing analgesia through additive or synergistic effects. The primary goal is generally to reduce or entirely eliminate the use of potent opioids, which are associated with numerous disadvantages and unacceptable side effects.

The American Pain Society (APS), in a guideline prepared by the American Society of Anesthesiologists (ASA), has recommended the implementation of multimodal analgesia in pain management strategies. The guideline strongly recommends, with high-quality evidence, that patients without contraindications receive paracetamol and/or nonsteroidal anti-inflammatory drugs (NSAIDs) as part of multimodal analgesia for postoperative pain management. It further indicates that paracetamol and NSAIDs possess different mechanisms of action, and their combination may be more effective than either drug alone. Additionally, the guideline advises clinicians to consider regional local anesthetic infiltration at the surgical site, supported by evidence of its efficacy (weak recommendation, moderate-quality evidence). The infiltration of long-acting local anesthetics in the surgical area has proven effective as a component of multimodal analgesia in various procedures.

Overall, research on multimodal analgesia has encountered difficulties in yielding consistent results due to variability in the types of analgesics used, their dosages, and drug combinations. Since some of these techniques are relatively new while others are still under development, further research is needed to fully ascertain the synergistic effects of multimodal analgesia strategies. Moreover, there is limited literature regarding the clinical efficacy of combinations involving three or more analgesics.

In light of these findings, there is a clear need for comprehensive research on multimodal analgesia strategies. Based on the recommendations of ERAS guidelines, this study was conceived to contribute to the literature by determining the synergistic analgesic efficacy achievable through the combination of different pain management mechanisms. Specifically, the efficacy of administering paracetamol and NSAIDs at appropriate times and dosages, along with the effectiveness of local anesthetic infiltration targeted at the surgical site for postoperative pain control, will be investigated. This study aims to evaluate the effects of ERAS protocol-based multimodal analgesia principles on postoperative pain, length of hospital stay, complications, and additional opioid requirements in patients undergoing laparoscopic cholecystectomy.

Methods

This non-randomized controlled study (an Ambispective Cohort Study) will be conducted on patients undergoing laparoscopic cholecystectomy in the general surgery clinic of a private hospital. The implementation of evidence-based ERAS protocols in the hospital has provided an opportunity to compare these protocols with the standard procedures performed previously. Thus, the study will involve prospectively observing patients managed according to the ERAS pain protocol (observation group) and retrospectively analyzing records of patients managed with the routine protocol before the implementation of ERAS (control group). The primary outcome is the evaluation of pain, while the secondary outcomes include hospital length of stay, early complication rates, and additional opioid requirements. The retrospective control group will consist of patients who received routine pain management in 2024, whereas the prospective observation group will consist of patients receiving the ERAS multimodal analgesia protocol between April and July 2025.

No premedication is administered to participants for sedation. Patients are routinely monitored in the operating room using standard procedures, including heart rate (HR), non-invasive blood pressure (NIBP), electrocardiogram (ECG), peripheral oxygen saturation (SpO₂), and body temperature monitoring with an esophageal probe. A standardized general anesthesia protocol is administered to all patients by an experienced anesthesiologist. Intravenous patient-controlled analgesia (IV PCA) is not used. After post-anesthesia care unit (PACU) monitoring, patients are transferred to the clinical ward. These procedures apply to both groups.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective laparoscopic cholecystectomy
* Classified as ASA (American Society of Anesthesiologists) class I-II

Exclusion Criteria:

* Patients with incomplete or insufficient medical records,
* Those undergoing concurrent major surgical procedures,
* Opioid users,
* ASA class III-IV patients,
* Those with hemorrhagic diathesis or coagulation disorders,
* A history of hypersensitivity to any medication used in this study
* Patients with peptic ulcer disease or gastrointestinal bleeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients treated with the ERAS multimodal analgesia protocol between 2024 and 2025 who were treated with the routine pain management protocol of 2024. The sample size was also determined by power analysis.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Pain levels will be measured | VAS score of pain at 2, 4, 8, 12, 18 and 24 hours in the recovery room and clinic
  Patients' pain will be measured with Visual Analog Scale (VAS) (0 to 10, where 0 = no pain and 10 = the worst imaginable pain). A score of 1-3 represents mild pain, 4-6 represents moderate pain, and 7-10 represents severe and unbearable pain .

SECONDARY OUTCOMES:
The length of hospital stay will be measured | Time interval from hospitalisation to discharge (assessed up to 5 days).
  The discharge date and time of the patients will be recorded and the duration of their hospital stay will be determined.
Total Additional Rate of Opioid Consumption During Hospital Stay | Time interval from the postoperative period until discharge (From postoperative Day 0 to postoperative Day 3)
  Rescue (additional) opioids used in the postoperative period will be determined.
Incidence of Early Postoperative Complications | Intraoperative and postoperative time interval (postoperative Day 5)
  Intraoperative events, postoperative adverse events will be recorded. In addition, postoperative complications will be determined according to the Clavien-Dindo classification system.

CONTACTS AND LOCATIONS:
Overall Officials: Esma Gökçe, Principal Investigator — Toros University
Locations (1):
- Cukurova University, Sarıçam, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nechay T, Titkova S, Tyagunov A, Anurov M, Sazhin A. Modified enhanced recovery after surgery protocol in patients with acute cholecystitis: efficacy, safety and feasibility. Multicenter randomized control study. Updates Surg. 2021 Aug;73(4):1407-1417. doi: 10.1007/s13304-021-01031-5. Epub 2021 Mar 22. PMID 33751409
- [Background] Yu T, Zhao L, Zhao H, Fu H, Li J, Yu A. The enhanced recovery after surgery (ERAS) protocol in elderly patients with acute cholecystitis: A retrospective study. Medicine (Baltimore). 2023 Feb 10;102(6):e32942. doi: 10.1097/MD.0000000000032942. PMID 36820555
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Gustafsson UO, Scott MJ, Hubner M, Nygren J, Demartines N, Francis N, Rockall TA, Young-Fadok TM, Hill AG, Soop M, de Boer HD, Urman RD, Chang GJ, Fichera A, Kessler H, Grass F, Whang EE, Fawcett WJ, Carli F, Lobo DN, Rollins KE, Balfour A, Baldini G, Riedel B, Ljungqvist O. Guidelines for Perioperative Care in Elective Colorectal Surgery: Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations: 2018. World J Surg. 2019 Mar;43(3):659-695. doi: 10.1007/s00268-018-4844-y. PMID 30426190
- [Background] Rawal N. Current issues in postoperative pain management. Eur J Anaesthesiol. 2016 Mar;33(3):160-71. doi: 10.1097/EJA.0000000000000366. PMID 26509324
- [Background] Wu CL, Raja SN. Treatment of acute postoperative pain. Lancet. 2011 Jun 25;377(9784):2215-25. doi: 10.1016/S0140-6736(11)60245-6. PMID 21704871
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Ong CK, Seymour RA, Lirk P, Merry AF. Combining paracetamol (acetaminophen) with nonsteroidal antiinflammatory drugs: a qualitative systematic review of analgesic efficacy for acute postoperative pain. Anesth Analg. 2010 Apr 1;110(4):1170-9. doi: 10.1213/ANE.0b013e3181cf9281. Epub 2010 Feb 8. PMID 20142348
- [Background] Kehlet H, Andersen LO. Local infiltration analgesia in joint replacement: the evidence and recommendations for clinical practice. Acta Anaesthesiol Scand. 2011 Aug;55(7):778-84. doi: 10.1111/j.1399-6576.2011.02429.x. Epub 2011 Apr 4. PMID 21463261
- [Background] Joshi GP, Schug SA, Kehlet H. Procedure-specific pain management and outcome strategies. Best Pract Res Clin Anaesthesiol. 2014 Jun;28(2):191-201. doi: 10.1016/j.bpa.2014.03.005. Epub 2014 May 9. PMID 24993439
- [Background] Nyundo M, Kayondo K, Gasakure M, Twagirumukiza JD, Gashegu J, Detry O. Implementation and outcomes of an enhanced recovery after surgery pathway for laparoscopic cholecystectomy in East and Central Africa: A prospective non-randomized controlled trial in Rwanda's Tertiary Teaching Hospital. World J Surg. 2025 Mar;49(3):605-614. doi: 10.1002/wjs.12371. Epub 2024 Oct 10. PMID 39390308
- [Background] Akbas S, Ozkan AS, Durak MA, Yologlu S. Efficacy of Intravenous Paracetamol and Ibuprofen on Postoperative Pain and Morphine Consumption in Lumbar Disc Surgery: Prospective, Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Neurochirurgie. 2021 Nov;67(6):533-539. doi: 10.1016/j.neuchi.2021.04.019. Epub 2021 May 11. PMID 33989641
- [Background] Freys JC, Bigalke SM, Mertes M, Lobo DN, Pogatzki-Zahn EM, Freys SM; PROSPECT Working Group of the European Society of Regional Anaesthesia and Pain Therapy (ESRA). Perioperative pain management for appendicectomy: A systematic review and Procedure-specific Postoperative Pain Management recommendations. Eur J Anaesthesiol. 2024 Mar 1;41(3):174-187. doi: 10.1097/EJA.0000000000001953. Epub 2024 Jan 12. PMID 38214556